CLINICAL TRIAL: NCT06991517
Title: A Prospective Cohort Study of Bicuspid Case Selection and Valve Sizing Using the ABC Bicuspid Sizing Algorithm for Sapien 3 Balloon Expandable Valve
Brief Title: A Study of Transcatheter Aortic Valve Replacement Case Selection and Valve Sizing Using the ABC Bicuspid Sizing Algorithm
Status: Recruiting | Type: Observational
Sponsor: World Health Research Inc. (Industry)
Collaborators: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Other Study IDs: 5168-CTIA-Feb/2025-117711
Record Dates: First submitted 2025-04-16; First posted 2025-05-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Aortic Stenosis
Keywords: Bicuspid Aortic Stenosis; Transcatheter Aortic Valve Replacement
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: The ABC Bicuspid Sizing Algorithm — The ABC Bicuspid Sizing Algorithm is a valve sizing algorithm. It guides operators' evaluations of CT scans, helping inform (1) treatment allocation between TAVR and surgical aortic valve replacement, and (2) valve choice for patients undergoing TAVR. In select cases, the algorithm will suggest gated CT evaluation or artificial intelligence-based simulation models be used to further evaluate the risk of the planned valve size and deployment volume. The operators will consider the findings of the ABC Bicuspid Sizing Algorithm as well as other clinical factors when making their final treatment decisions.

SUMMARY:
The goal of this study is to learn what effects the ABC Bicuspid Sizing Algorithm has on the clinical outcomes of patients with bicuspid aortic stenosis after having a transcatheter aortic valve replacement (TAVR) using the Sapien 3 valve. The main questions the study aims to answer are:

1. Does the ABC Bicuspid Sizing Algorithm increase the technical success at exit from the procedure room?
2. Does the ABC Bicuspid Sizing Algorithm increase the device success at 30 days after the procedure?

Participants already being evaluated for a TAVR as part of their regular medical care for bicuspid aortic stenosis will have their diagnostic images assessed using the ABC Bicuspid Sizing Algorithm to help determine their procedure type and valve size. They will have visits 30 days and one year after their procedure.

DETAILED DESCRIPTION:
This is a multi-centre, international, prospective cohort study. Approximately 290 patients who are clinically eligible for transcatheter aortic valve replacement (TAVR) will be enrolled. Using information collected with the ABC Bicuspid Sizing Algorithm, physicians will make a treatment allocation between TAVR and surgical aortic valve replacement (SAVR), and determine valve sizing and deployment for TAVR-treated patients. Included in the algorithm use is the utilization of gated computed tomography evaluation or artificial intelligence-based simulation models in select cases with borderline feasibility. The findings of these additional assessments will be shared with the treating physicians for consideration in the final treatment decision.

Of the 290 patients, an estimated 230 will be recommended to have TAVR. Data will be collected from TAVR-treated patients at baseline, procedure, hospital discharge, and 30 days and one year after the procedure. Data will only be collected from SAVR-treated patients at baseline and procedure. Sites in Canada, Latin America, the Middle East, and Asia Pacific will participate.

ELIGIBILITY:
Inclusion Criteria:

* Have bicuspid aortic valve disease
* Have severe aortic stenosis or mixed aortic stenosis and regurgitation requiring treatment
* Have no other condition requiring surgical intervention
* Have had a TAVR CT scan (retrospectively gated contrast enhanced acquisition) that is of diagnostic quality and includes multiphase reconstructions of the aortic root at the minimum available slice thickness (with at least three systolic and one diastolic phases)
* Would be treated with a Sapien 3 valve if found to be anatomically suitable for TAVR
* Have a suitable access route for TAVR with a Sapien 3 valve

Exclusion Criteria:

* Are treated with TAVR using a device other than a Sapien 3 valve
* Are unable to be treated with TAVR due to intercurrent illness, clinical instability, or death on waitlist after being accepted for TAVR

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients referred to the TAVR program at select hospitals
Sampling Method: Non-Probability Sample
Enrollment: 290 (Estimated)
Dates: Start 2025-05-13 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of cases achieving technical success | At exit from procedure room after procedure completion
  Freedom from mortality, successful access, delivery of the device, and retrieval of the delivery system, correct positioning of a single prosthetic heart valve into the proper anatomical location, and freedom from surgery or intervention related to the device or cardiac structural complication

SECONDARY OUTCOMES:
Proportion of cases achieving device success | At 30 days after the procedure
  Technical success and intended performance of the valve (mean gradient less than 20 mmHg, peak velocity less than 3 m/s, Doppler velocity index greater than 0.35, and less than moderate aortic regurgitation)
Proportion of cases in which the use of gated computed tomography evaluation or artificial intelligence-based simulation models altered the treatment plan or operator confidence in the treatment plan compared to the ABC Bicuspid Sizing Algorithm alone | At baseline
New conduction disturbance and permanent pacemaker implantation | At 30 days and 1 year after the procedure
Stroke or transient ischemic attack | At 30 days and 1 year after the procedure
Major vascular complication | At 30 days after the procedure
Moderate or severe paravalvular regurgitation | At 30 days and 1 year after the procedure
Death | At 30 days and 1 year after the procedure
Acute valve complication | At 30 days and 1 year after the procedure
Need for cardiac surgery | At 30 days and 1 year after the procedure
Delayed valve dysfunction | At 1 year after the procedure
Proportion of cases in which evaluation of anatomy above or below the annulus altered the valve sizing and deployment decision compared to the calculated valve sizing and deployment decision considering the annulus size only | At baseline

CONTACTS AND LOCATIONS:
Overall Officials: Tej PM Sheth, MD, FRCPC, Principal Investigator — McMaster University, World Health Research Inc.
Locations (21):
- Australia (7):
  - John Hunter Hospital, New Lambton Heights, New South Wales
  - North Shore Private Hospital, St Leonards, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - The Prince Charles Hospital, Chermside, Queensland
  - St Andrew's War Memorial Hospital, Spring Hill, Queensland
  - The Alfred, Melbourne, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
- Canada (7):
  - Foothills Medical Centre, Calgary, Alberta
  - NovaScotia Health Authority- Halifax Infimary, Halifax, NovaScotia
  - Hamilton General Hospital, Hamilton, Ontario
  - Southlake Regional Health Centre, Newmarket, Ontario
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Institut universitaire de cardiologie et de pneumologie de Québec - Université Laval, Québec, Quebec
- Fundación Cardioinfantil - LaCardio, Bogotá, Colombia
- Hospital San Juan de Dios, San José, Provincia de San José, Costa Rica
- Mexico (2):
  - Centro Médico Nacional Siglo XXI, Mexico City
  - Instituto Nacional de Cardiología - Ignacio Chávez, Mexico City
- Wellington Regional Hospital, Newtown, Wellington Region, New Zealand
- National Heart Centre Singapore, Singapore, Singapore
- Ramathibodi Hospital, Bangkok, Thailand